CLINICAL TRIAL: NCT02977936
Title: Descriptive Study for the Management of Joint Pain Associated With Osteoarthritis of the Knee: Association of Extracts of Curcuma Longa, Boswellia Serrata and Porphyra Umbilicalis.
Brief Title: Management of Joint Pain Associated With Osteoarthritis of the Knee With Association of Plant Extracts.
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PiL-Obs-CFort-016
Record Dates: First submitted 2016-11-25; First posted 2016-11-30 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Cartimotil Fort — 1 to 4 capsules per day during 90 days

SUMMARY:
The aim of the study is to evaluate at 3 months the effect of a supplementation with extracts of Curcuma longa, Boswellia serrata and Porphyra umbilicalis on the acceptability of pain for patients suffering from gonarthritic pain.

DETAILED DESCRIPTION:
For this study, 126 patients are going to be included. They will have a supplementation of Cartimotil Fort®, from 1 to 4 capsules per day during 90 days.

on the one hand, during the two visits (inclusion and follow-up), the investigator completes the questionnaire about neuropathic pain (DN4).

on the other hand, patients complete the Osteoarthritis Symptom Inventory Scale (OASIS) 4 times : just after the inclusion visit, at day 30, at day 60 and just before the follow-up visit (day 90). He completes the Patient Global Impression of Improvement (PGII), the Minimal Clinically Important Improvement (MCII) and the Acceptable Symptomatic Statement (PASS) 6 times : just after the inclusion visit, at day 10, at day 20, at day 30, at day 60 and just before the follow-up visit (day 90).

ELIGIBILITY:
Inclusion Criteria:

* VAS of pain : minimum 5/10 on walking or 4/10 at rest
* Patients with a negative PASS (patient considering that the symptomatic state is not acceptable)
* Suffering from mono or bilateral femoro-tibial knee osteoarthrosis with painful seizures (confirmed by a radio of less than two years: stage 2 or 3 on the Kellgreen scale - clinical examination)
* Having agreed to participate in the investigation after receiving information from the investigator

Exclusion Criteria:

* Patients with rheumatological disorders other than osteoarthritis
* Patients for whom knee surgery is planned within 3 months
* Patients who started treatment with chondroitin sulphate (or all treatments of osteoarthritis other than anti-inflammatories and analgesics) for less than one month
* Patients with a BMI greater than 35
* Patients with chronic pain that can interfere with knee osteoarthritis pain
* Patients with reduced mobility or bedridden
* Patients with cognitive impairments not able to participate in the study
* Patients with known allergies to any of the ingredients of Cartimotil Fort®
* Pregnant or breastfeeding patients
* Patients who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from gonarthrosic pain
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching the acceptability threshold of their state | day 30
  Percentage of patients reaching the acceptability threshold of their state between D0 and D30 measured by the binary response of the PASS (yes = acceptable).

SECONDARY OUTCOMES:
OASIS Score | Day 30
OASIS Score | Day 60
OASIS Score | Day 90
Yes answer for the PASS | Day 60
Yes answer for the PASS | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Pileje Network of medical practitioners in private offices, Paris, France

REFERENCES:
- [Derived] Perrot S, Trouvin AP, Bouhassira D. Three dimensions of pain in osteoarthritis: development and validation of the Osteoarthritis Symptom Inventory Scale. Pain. 2023 Jul 1;164(7):1566-1577. doi: 10.1097/j.pain.0000000000002856. Epub 2023 Mar 22. PMID 36602324